CLINICAL TRIAL: NCT00310713
Title: A Phase IV, Single Centre, Open-label Study to Investigate the Kinetics of the B Cell Response to the C Saccharide Component of Chiron's Meningococcal C Conjugate Vaccine Administered to Healthy Children at Least 12 Months of Age After Priming With a Commercially Available Men ACWY Conjugate Vaccine at 2, 3 and 4 Months of Age
Brief Title: Persistence of Antibodies and Kinetics of B Cell Response in Healthy Children After Vaccination With MCC Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: M14P5E1; Impact N° 1637
Record Dates: First submitted 2006-04-03; First posted 2006-04-04 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Prevention of Meningococcal Infection
Keywords: Prevention of Meningococcal Meningitis; vaccines; conjugate; immunology; children; antibody persistence
MeSH Terms: interventions — serogroup C meningococcal conjugate vaccine

ARMS (5):
- Group 1 (Experimental)
  Interventions: Biological: Meningococcal C conjugate vaccine
- Group 2 (Experimental)
  Interventions: Biological: Meningococcal C conjugate vaccine
- Group 3 (Experimental)
  Interventions: Biological: Meningococcal C conjugate vaccine
- Group 4 (Experimental)
  Interventions: Biological: Meningococcal C conjugate vaccine
- Group 5 (Experimental)
  Interventions: Biological: Meningococcal C conjugate vaccine

INTERVENTIONS:
Biological: Meningococcal C conjugate vaccine — Group 1: Meningococcal C conjugate vaccine dose boost on Visit 6 (day 0), blood sample on Visit 7 (day 3 post immunization) Group 2: Meningococcal C conjugate vaccine dose boost on Visit 6 (day 0), blood sample on Visit 7 (day 5 post immunization) Group 3: Meningococcal C conjugate vaccine dose boost on Visit 6 (day 0), blood sample on Visit 7 (day 7 post immunization) Group 4: Meningococcal C conjugate vaccine dose boost on Visit 6 (day 0), blood sample on Visit 7 (day 9 post immunization) Group 5: Meningococcal C conjugate vaccine dose boost on Visit 6 (day 0), blood sample on Visit 7 (day 10 post immunization)

SUMMARY:
Persistence of antibodies and kinetics of B cell response in healthy children after vaccination with MCC vaccine

ELIGIBILITY:
Inclusion Criteria:

* Healthy children

Exclusion Criteria:

* Known hypersensitivity to any vaccine products
* Any immunodeficiency, genetic anomaly or severe acute or chronic illness

Ages: 12 Months to 13 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2006-04; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Persistence of memory B cells in the blood at least one year after primary immunisation with MenC Vaccine at 2, 3 and 4 months of age, as determined by meningococcal C specific B-cell ELISPot assay or limiting dilution

SECONDARY OUTCOMES:
Immune Response measured 4 weeks after the booster immunisation.
establish at which day CRM -197 specific B cells are detectable in the blood after booster immunisation, as determined by meningococcal C specific B-cell ELISpot assay or limiting dilution.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines - Information Services, Principal Investigator — Novartis Vaccines & Diagnostics
Locations (1):
- Oxford Vaccine Group, Centre for Clinical Vaccinology and Tropical Medicine, Churchill Hospital, Old Road, Headington, Oxford, United Kingdom

REFERENCES:
- [Background] Blanchard Rohner G, Snape MD, Kelly DF, John T, Morant A, Yu LM, Borkowski A, Ceddia F, Borrow R, Siegrist CA, Pollard AJ. The magnitude of the antibody and memory B cell responses during priming with a protein-polysaccharide conjugate vaccine in human infants is associated with the persistence of antibody and the intensity of booster response. J Immunol. 2008 Feb 15;180(4):2165-73. doi: 10.4049/jimmunol.180.4.2165. PMID 18250423